CLINICAL TRIAL: NCT00574704
Title: Double Blind Placebo Controlled Study to Assess Efficacy and Safety of a Combined Allergen Vaccine (CYT005-AllQbG10) and Its Single Components in Patients With House Dust Mite Allergy
Brief Title: A Study to Investigate an Immunomodulatory Therapy in Adult Patients With Perennial Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT005-AllQbG10 03
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-02

CONDITIONS: Perennial Allergic Rhinoconjunctivitis; House Dust Mite Allergy
MeSH Terms: conditions — Dust Mite Allergy | interventions — CYT003-QbG10; Antigens, Dermatophagoides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: CYT005-AllQbG10 (combination of house dust mite allergen extract with CYT003-QbG10)
- 2 (Placebo Comparator)
  Interventions: Drug: House dust mite allergen extract in combination with CYT003-QbG10-placebo
- 3 (Experimental)
  Interventions: Drug: CYT003-AllQbG10 in combination with house dust mite allergen extract placebo
- 4 (Placebo Comparator)
  Interventions: Drug: CYT003-QbG10-placebo in combination with house dust mite allergen extract placebo

INTERVENTIONS:
Drug: CYT005-AllQbG10 (combination of house dust mite allergen extract with CYT003-QbG10) — subcutaneous injections at 6 visits
  Arms: 1
Drug: House dust mite allergen extract in combination with CYT003-QbG10-placebo — subcutaneous injections at 6 visits
  Arms: 2
Drug: CYT003-AllQbG10 in combination with house dust mite allergen extract placebo — subcutaneous injections at 6 visits
  Arms: 3
Drug: CYT003-QbG10-placebo in combination with house dust mite allergen extract placebo — subcutaneous injections at 6 visits
  Arms: 4

SUMMARY:
The purpose of the study is to test the efficacy of the combination treatment AllQbG10 in patients with perennial allergic rhinoconjunctivitis due to house dust mite allergy in a double-blind, placebo-controlled setting

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate perennial allergic rhinoconjunctivitis due to hypersensitization towards house dust mite allergens

Exclusion Criteria:

* Clinically relevant other allergies (perennial or seasonal) that could potentially interfere with the patient's study treatment schedule or assessments
* Use of any concomitant medication that could affect the patient's study treatment response or assessment results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Mueller, MD, Study Director — Cytos Biotechnology

RESULTS

PARTICIPANT FLOW:
Groups:
- AllQbG10: CYT005-AllQbG10 (combination of house dust mite allergen extract with CYT003-QbG10) : subcutaneous injections at 6 visits
- Allergen: House dust mite allergen extract in combination with CYT003-QbG10-placebo : subcutaneous injections at 6 visits
- QbG10: CYT003-AllQbG10 in combination with house dust mite allergen extract placebo : subcutaneous injections at 6 visits
- Placebo: CYT003-QbG10-placebo in combination with house dust mite allergen extract placebo : subcutaneous injections at 6 visits
Period: Overall Study
Arm/Group | AllQbG10 | Allergen | QbG10 | Placebo
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 9 | 10
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AllQbG10 | Allergen | QbG10 | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.2 (8.6) | 36.5 (9.8) | 36.8 (11.0) | 31.0 (15.9) | 34.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 4 | 16
  Male | 7 | 4 | 7 | 6 | 24
Region of Enrollment [Number; unit: participants]
  Europe | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Provocation Test (CPT) With House Dust Mite Allergen Solutions. Change of Median Individual Allergen Tolerance Compared to Baseline (Factor of Increase in Allergen Concentration to Induce a Threshold CPT Score ≥ 2)
Description: The outcome measure is a conjunctival provocation test (CPT) with house dust mite allergen solutions. CPT score was measured as a sum of the following assessed symptoms: conjunctival hyperemia, tearing, itching, burning and swelling of eyelids. Each of the assessed symptom could be absent (0), mild (1 point), moderate (2 points) or severe (3 points). The provocation tests started with the maximal dilution of the allergen 1:1000. If the sum of the reached CPT score was <10 points, the test continued with the next dilution step 1:100. This procedure was repeated until patients reached the CPT score ≥ 10 points or the provocation solution reached the maximal concentration 1:1 (undiluted).
  The outcome is then given as the change of median individual allergen tolerance at month two compared to baseline. The change is expressed as a factor of increase in allergen concentration to induce a threshold CPT score ≥ 2.
Time Frame: baseline versus 2 months after baseline
Measure: Median (Inter-Quartile Range); unit: Factor of Increased Allergen Tolerance
Arm/Group | AllQbG10 | Allergen | QbG10 | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Factor of Increased Allergen Tolerance | 10 [1.0 to 100.0] | 10 [1.0 to 10.0] | 10 [1.0 to 10.0] | 1 [0.1 to 10.0]

2. Secondary Outcome: Safety and Tolerability of the Study Treatment by Collection of Adverse Events
Time Frame: about 30 min. at each visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | AllQbG10 | Allergen | QbG10 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 10/10 | 8/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AllQbG10 (N=10) | Allergen (N=10) | QbG10 (N=10) | Placebo (N=10)
fracture of right malleolus (accident) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AllQbG10 (N=10) | Allergen (N=10) | QbG10 (N=10) | Placebo (N=10)
Nasopharyngitis (Infections and infestations) | 4 | 1 | 4 | 5
Influenza (Infections and infestations) | 3 | 3 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 2 | 1 | 2
Local reactions (General disorders) | 2 | 2 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days